CLINICAL TRIAL: NCT05907395
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, 4-PERIOD, CROSSOVER, FIRST-IN-HUMAN STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING ORAL DOSES OF PF-07293893 ADMINISTERED TO HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About the Study Medicine (PF-07293893) at Different Dose Levels in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C5171001; 2023-504921-37-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: PF-07293893; Single ascending dose; Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PF-07293893 and Placebo (Cohort 1) (Experimental): Single dose administration of PF-07293893 and placebo; Within a cohort, participants will receive up to 4 doses of PF-07293893 and up to 2 doses of placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 2) (Experimental): Single dose administration of PF-07293893 and placebo; Within a cohort, participants will receive up to 4 doses of PF-07293893 and up to 2 doses of placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 3) (Experimental): Single dose administration of PF-07293893 and placebo; Within a cohort, participants will receive up to 4 doses of PF-07293893 and up to 2 doses of placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo

INTERVENTIONS:
Drug: PF-07293893 — PF-07293893 will be prepared as an oral suspension given in escalating single doses to be determined.
Drug: Placebo — Matching placebo will be prepared as an oral suspension given in each cohort.

SUMMARY:
The purposes of the study are:

To learn about the safety and tolerability of study medicine (PF-07293893). Tolerability is the extent to which side effects can be tolerated. Side effects are unwanted reactions to the study medicine.

To measure the amount of PF-07293893 in blood after the medicine is taken by mouth.

The study is seeking participants who:

* Are females of non-childbearing potential and males 18 to 65 years of age
* Are in generally healthy condition
* Have not had viral infections (HIV, HBV or HCV). HIV, human immunodeficiency virus. HBV, human hepatitis B virus. HCV, human hepatitis C virus.

Participants will receive either PF-07293893 or placebo (dummy pill) by chance. Participants will undergo up to 4 treatments periods in this study. Everyone will receive up to 4 doses of study medicine and up to 2 doses of placebo. In each period, participants will stay in study clinic for 5 days. There will be at least 2 days between each treatment period.

Participants will be involved in this study for about 14 weeks. During their stay, participants will undergo several examinations. Participants will also have their blood collected by the study doctors for several times.

ELIGIBILITY:
This study is seeking participants who are:

* Females of non-childbearing potential and males 18 to 65 years of age, inclusive, at the time of signing the informed consent document (ICD) who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

This study is not seeking participants who have:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* History of human immunodeficiency virus infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen, or hepatitis C antibody. Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to coronavirus disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest.
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR) <75 mL/min/1.73m².
* Standard 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin ≥1.05 × upper limit of normal (ULN), participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5171001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 participants (initially randomized participants and replacement participants) were enrolled in this study. All participants received at least 1 dose of study intervention and were assigned in the study into 3 cohorts. As planned, there were "replacement" participants in the study who were not initially randomized, but they replaced those participants who discontinued in any treatment period due to reasons other than safety; this was per investigator's and sponsor's discretion.
Groups:
- Cohort 1: Sequence 1: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 10 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 30 mg; then Period 3/Day1 (SDD, fasted): PF-07293893 100 mg; then Period 4/Day1 (SDD, fasted): placebo matched to PF-07293893. SDD = spray dried dispersion form.
- Cohort 1: Sequence 2: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 10 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 30 mg; then Period 3/Day1 (SDD, fasted): placebo matched to PF-07293893; then Period 4/Day1 (SDD, fasted): PF-07293893 300 mg.
- Cohort 1: Sequence 3: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 10 mg; then Period 2/Day 1 (SDD, fasted): placebo matched to PF-07293893; then Period 3/Day1 (SDD, fasted): PF-07293893 100 mg; then Period 4/Day1 (SDD, fasted): PF-07293893 300 mg.
- Cohort 1: Sequence 4: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): placebo matched to PF-07293893; then Period 2/Day 1 (SDD, fasted): PF-07293893 30 mg; then Period 3/Day1 (SDD, fasted): PF-07293893 100 mg; then Period 4/Day1 (SDD, fasted): PF-07293893 300 mg.
- Cohort 2: Sequence 1: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 1500 mg; then Period 3/Day1 (CRYS, fasted): PF-07293893 300 mg; then Period 4/Day1 (CRYS, fed): PF-07293893 300 mg. CRYS = crystalline form.
- Cohort 2: Sequence 2: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 1500 mg; then Period 3/Day1 (CRYS, fasted): placebo matched to PF-07293893; then Period 4/Day1 (CRYS, fed): placebo matched to PF-07293893.
- Cohort 2: Sequence 3: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): placebo matched to PF-07293893; then Period 3/Day1 (CRYS, fasted):PF-07293893 300 mg; then Period 4/Day1 (CRYS, fed): PF-07293893 300 mg.
- Cohort 2: Sequence 4: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fasted): placebo matched to PF-07293893; then Period 2/Day 1 (SDD, fasted): PF 07293893 1500 mg; then Period 3/Day1 (CRYS, fasted): PF-07293893 300 mg; then Period 4/Day1 (CRYS, fed): PF-07293893 300 mg.
- Cohort 3: Sequence 1: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fed): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 1200 mg; then Period 3/Day1 (SDD, fasted): PF-07293893 900 mg; then Period 4/Day1 (SDD, fasted): PF-07293893 750 mg.
- Cohort 3: Sequence 2: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fed): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): PF-07293893 1200 mg; then Period 3/Day1 (SDD, fasted): placebo matched to PF-07293893; then Period 4/Day1 (SDD, fasted): PF-07293893 750 mg.
- Cohort 3: Sequence 3: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fed): PF-07293893 750 mg; then Period 2/Day 1 (SDD, fasted): placebo matched to PF-07293893; then Period 3/Day1 (SDD, fasted): PF-07293893 900 mg; then Period 4/Day1 (SDD, fasted): PF-07293893 750 mg.
- Cohort 3: Sequence 4: Participants received treatment as oral suspension in all periods. Period 1/Day1 (SDD, fed): placebo matched to PF-07293893; then Period 2/Day 1 (SDD, fasted): PF-07293893 1200 mg; then Period 3/Day1 (SDD, fasted): PF-07293893 900 mg; then Period 4/Day1 (SDD, fasted): placebo matched to PF-07293893.
Period: Period 1
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3 | Cohort 3: Sequence 4
Started (Participants who entered period 1.) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3 | Cohort 3: Sequence 4
Started (Participants who entered period 2.) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Personal reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3 | Cohort 3: Sequence 4
Started (Participants who entered period 3.) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 1: Sequence 4 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4 | Cohort 3: Sequence 1 | Cohort 3: Sequence 2 | Cohort 3: Sequence 3 | Cohort 3: Sequence 4
Started (Participants who entered period 4.) | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Except the replacement participants, all participants were randomized to receive all interventions in a cohort. Thus, the participants in a cohort were combined in the record.
Groups:
- Cohort 1: In this cohort participants were randomized to received placebo matched to PF-07293893 or PF-07293893 (10 mg, 30 mg, 100 mg or 300 mg) in sequence 1 or 2 or 3 or 4.
- Cohort 2: In this cohort participants were randomized to received placebo matched to PF-07293893 or PF-07293893 (300mg [fast/fed],750 mg, 1500 mg) in sequence 1 or 2 or 3 or 4.
- Cohort 3: In this cohort participants were randomized to received placebo matched to PF-07293893 or PF-07293893 (750 mg [fast/fed], 900 mg, 1200 mg) in sequence 1 or 2 or 3 or 4.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 10 | 11 | 9 | 30
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-44 Years | 6 | 7 | 4 | 17
  Age: 45-64 Years | 4 | 4 | 4 | 12
  Age: >=65 Years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 11 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 10 | 8 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were events with onset dates on or after the start of the study drug.
Time Frame: Day 1 of first dose up to maximum of 35 days post last dose (up to 60 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- PF-07293893 10 mg: SDD/Fasted Cohort 1: Participants received PF-07293893 SDD 10 mg in fasted condition.
- PF-07293893 30 mg: SDD/Fasted Cohort 1: Participants received PF-07293893 SDD 30 mg in fasted condition.
- PF-07293893 100 mg: SDD/Fasted Cohort 1: Participants received PF-07293893 SDD100 mg in fasted condition.
- PF-07293893 300 mg: CRYS/Fasted Cohort 2: Participants received PF-07293893 CRYS 300 mg in fasted condition.
- PF-07293893 300 mg: CRYS/Fed Cohort 2: Participants received PF-07293893 CRYS 300 mg in fed condition.
- PF-07293893 300 mg: SDD/Fasted Cohort 1: Participants received PF-07293893 SDD 300 mg in fasted condition.
- PF-07293893 750 mg: SDD/Fasted Cohort 2; PF-07293893 750 mg: SDD/Fasted Cohort 3: Participants received PF-07293893 SDD 750 mg in fasted condition.
- PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3: Participants who received PF-07293893 SDD 750 mg in fasted condition.
- PF-07293893 750 mg: SDD/Fed Cohort 3: Participants received PF-07293893 SDD 750 mg in fed condition.
- PF-07293893 900 mg: SDD/Fasted Cohort 3: Participants received PF-07293893 SDD 900 mg in fasted condition.
- PF-07293893 1200 mg: SDD/Fasted Cohort 3: Participants received PF-07293893 SDD 1200 mg in fasted condition.
- PF-07293893 1500 mg: SDD/Fasted Cohort 2: Participants received PF-07293893 SDD 1500 mg in fasted condition.
- Placebo: CRYS/Fasted Cohort 2: Participants received placebo matched to PF-07293893 CRYS in fasted condition.
- Placebo: CRYS/Fed Cohort 2: Participants received placebo matched to PF-07293893 CRYS in fed condition.
- Placebo: SDD/Fasted Combined for All Cohorts: Participants received placebo matched to PF-07293893 SDD in fasted condition.
- Placebo: SDD/Fed Cohort 2: Participants received placebo matched to PF-07293893 SDD in fed condition.
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2 | Placebo: CRYS/Fasted Cohort 2 | Placebo: CRYS/Fed Cohort 2 | Placebo: SDD/Fasted Combined for All Cohorts | Placebo: SDD/Fed Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 2 | 2 | 18 | 2
Participants | 1 | 2 | 1 | 2 | 3 | 3 | 3 | 5 | 8 | 2 | 4 | 3 | 4 | 2 | 1 | 6 | 1

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Following parameters were analyzed for laboratory abnormalities: hematology (lymphocytes <0.8*lower limit of normal [LLN], lymphocytes/leukocytes <0.8*LLN, neutrophils <0.8*LLN, neutrophils/leukocytes <0.8*LLN, eosinophils/leukocytes >1.2*upper limit of normal [ULN], monocytes >1.2*ULN, monocytes/leukocytes >1.2*ULN); clinical chemistry (aspartate aminotransferase >3.0*ULN, potassium >1.1*ULN, creatine kinase >2.0*ULN); urinalysis (urine specific gravity <1.003 ,>1.030, ketones >=1, urine hemoglobin >=1, urobilinogen >=1, urine bilirubin >=1, leukocyte esterase >=1). In this outcome measure, participants with any laboratory abnormalities are reported.
Time Frame: Day 1 of first dose up to maximum of 9 days post last dose (up to 34 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2 | Placebo: CRYS/Fasted Cohort 2 | Placebo: CRYS/Fed Cohort 2 | Placebo: SDD/Fasted Combined for All Cohorts | Placebo: SDD/Fed Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 2 | 2 | 18 | 2
Participants | 3 | 3 | 4 | 2 | 2 | 2 | 1 | 2 | 3 | 4 | 4 | 3 | 3 | 2 | 1 | 7 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs assessments included blood pressure, pulse rate, respiratory rate and body temperature. Clinical significance of vital signs was determined based by investigator's discretion.
Time Frame: Day 1 of first dose up to maximum of 9 days post last dose (up to 34 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2 | Placebo: CRYS/Fasted Cohort 2 | Placebo: CRYS/Fed Cohort 2 | Placebo: SDD/Fasted Combined for All Cohorts | Placebo: SDD/Fed Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 2 | 2 | 18 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings
Description: ECG parameters included heart rate, PR interval, QTc corrected using Fridericia's formula (QTcF) and QRS complex. Clinically significant ECG findings were determined by the investigator's discretion.
Time Frame: Day 1 of first dose up to maximum of 9 days post last dose (up to 34 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2 | Placebo: CRYS/Fasted Cohort 2 | Placebo: CRYS/Fed Cohort 2 | Placebo: SDD/Fasted Combined for All Cohorts | Placebo: SDD/Fed Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 2 | 2 | 18 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-07293893
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24, 48 and 72 hours post dose of any treatment period
Population: Pharmacokinetic (PK) parameter Set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ mL)
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/ mL) | 110.2 (39) | 360.1 (19) | 1173 (24) | 147.2 (20) | 690.6 (23) | 3613 (34) | 5632 (28) | 6831 (9) | 6203 (22) | 5653 (33) | 7894 (15) | 7458 (18) | 7398 (22)

6. Secondary Outcome: Time for Cmax (Tmax) of PF-07293893
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24, 48 and 72 hours post dose of any treatment period
Population: PK parameter Set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated.
Measure: Median (Full Range); unit: Hour
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Hour | 1.00 [1.00 to 1.03] | 1.01 [1.00 to 1.03] | 2.03 [1.00 to 3.00] | 2.50 [1.00 to 4.03] | 6.00 [4.00 to 8.00] | 2.51 [2.00 to 3.00] | 3.51 [2.00 to 4.00] | 2.50 [1.00 to 6.22] | 3.01 [1.00 to 6.22] | 5.00 [4.00 to 6.00] | 4.00 [3.00 to 6.00] | 4.00 [3.00 to 6.03] | 4.01 [3.00 to 6.00]

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-07293893
Description: AUClast was calculated using linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24, 48 and 72 hours post dose of any treatment period
Population: PK Parameter Set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention and have at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/ mL)
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/ mL) | 782.5 (37) | 2671 (11) | 8354 (24) | 2057 (19) | 8910 (30) | 29900 (25) | 50150 (37) | 89220 (17) | 66890 (42) | 80700 (48) | 100700 (20) | 103400 (30) | 94210 (34)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07293893
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24, 48 and 72 hours post dose of any treatment period
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/ mL)
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/ mL) | 799.3 (36) | 2700 (11) | 8397 (24) | 2219 (20) | 9001 (30) | 30010 (25) | 50280 (37) | 89780 (17) | 67190 (42) | 81070 (49) | 101200 (21) | 103900 (30) | 94570 (34)

9. Secondary Outcome: Terminal Half-Life (t1/2) of PF-07293893
Description: t1/2 was calculated as log^e (2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24, 48 and 72 hours post dose of any treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Hour | 13.88 (2.8160) | 15.32 (1.4386) | 13.92 (2.0673) | 21.50 (6.5593) | 13.70 (1.2767) | 11.34 (2.1157) | 10.07 (3.0057) | 11.00 (1.3977) | 10.54 (2.2872) | 10.90 (1.2152) | 10.76 (1.3132) | 10.44 (2.1452) | 9.578 (1.1218)

ADVERSE EVENTS:
Time Frame: Day 1 of first dose up to maximum of 35 days post last dose (up to 60 days)
Arm/Group | PF-07293893 10 mg: SDD/Fasted Cohort 1 | PF-07293893 30 mg: SDD/Fasted Cohort 1 | PF-07293893 100 mg: SDD/Fasted Cohort 1 | PF-07293893 300 mg: CRYS/Fasted Cohort 2 | PF-07293893 300 mg: CRYS/Fed Cohort 2 | PF-07293893 300 mg: SDD/Fasted Cohort 1 | PF-07293893 750 mg: SDD/Fasted Cohort 2 | PF-07293893 750 mg: SDD/Fasted Cohort 3 | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 | PF-07293893 750 mg: SDD/Fed Cohort 3 | PF-07293893 900 mg: SDD/Fasted Cohort 3 | PF-07293893 1200 mg: SDD/Fasted Cohort 3 | PF-07293893 1500 mg: SDD/Fasted Cohort 2 | Placebo: CRYS/Fasted Cohort 2 | Placebo: CRYS/Fed Cohort 2 | Placebo: SDD/Fasted Combined for All Cohorts | Placebo: SDD/Fed Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/2 | 0/18 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/2 | 0/18 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/6 | 2/6 | 3/5 | 3/6 | 3/6 | 5/6 | 8/12 | 2/6 | 4/6 | 3/6 | 4/6 | 2/2 | 1/2 | 6/18 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07293893 10 mg: SDD/Fasted Cohort 1 (N=6) | PF-07293893 30 mg: SDD/Fasted Cohort 1 (N=6) | PF-07293893 100 mg: SDD/Fasted Cohort 1 (N=6) | PF-07293893 300 mg: CRYS/Fasted Cohort 2 (N=6) | PF-07293893 300 mg: CRYS/Fed Cohort 2 (N=5) | PF-07293893 300 mg: SDD/Fasted Cohort 1 (N=6) | PF-07293893 750 mg: SDD/Fasted Cohort 2 (N=6) | PF-07293893 750 mg: SDD/Fasted Cohort 3 (N=6) | PF-07293893 750 mg: SDD/Fasted Combined for Cohorts 2 and 3 (N=12) | PF-07293893 750 mg: SDD/Fed Cohort 3 (N=6) | PF-07293893 900 mg: SDD/Fasted Cohort 3 (N=6) | PF-07293893 1200 mg: SDD/Fasted Cohort 3 (N=6) | PF-07293893 1500 mg: SDD/Fasted Cohort 2 (N=6) | Placebo: CRYS/Fasted Cohort 2 (N=2) | Placebo: CRYS/Fed Cohort 2 (N=2) | Placebo: SDD/Fasted Combined for All Cohorts (N=18) | Placebo: SDD/Fed Cohort 2 (N=2)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4 | 6 | 1 | 2 | 2 | 4 | 1 | 1 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Any untoward findings identified on physical and/or neurological examinations, cardiac monitoring conducted during the active collection period were captured as adverse events, if those findings met the definition of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05907395/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05907395/SAP_001.pdf